CLINICAL TRIAL: NCT01927874
Title: Comparative Study of the Analgesic Effect of Subarachnoid or Infiltration for Hemorrhoidectomy
Brief Title: Subarachnoid or Infiltration for Hemorrhoidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rioko Kimiko Sakata, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bl.Pud
Record Dates: First submitted 2012-08-23; First posted 2013-08-23 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Hemorrhoid
Keywords: infiltration; hemorrhoidectomy; Postoperative pain
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative | interventions — Anesthesia, Local; Anesthesia, Spinal; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infiltration, analgesic effect (Active Comparator): 10ml 0.5% bupivacaine each side Block Injection of local anesthetic at pudendal nerve
  Interventions: Procedure: Infiltration; Drug: Bupivacaine
- Spinal block (Active Comparator): 10 mg of hyperbaric 0.5% bupivacaine Injection of anesthetic at subarachnoidal space
  Interventions: Procedure: Spinal block; Drug: 10 mg of hyperbaric 0.5% bupivacaine

INTERVENTIONS:
Procedure: Infiltration — injection of local anesthetic, associated with general anesthesia
  Other Names: Local Infiltration
  Arms: Infiltration, analgesic effect
Procedure: Spinal block — injection of anesthetic
  Other Names: subarachnoidal block
  Arms: Spinal block
Drug: Bupivacaine — 10ml 0.5% bupivacaine.
  Other Names: Local infiltration
  Arms: Infiltration, analgesic effect
Drug: 10 mg of hyperbaric 0.5% bupivacaine — Spinal punction and injection of local anesthetic
  Other Names: spinal anesthesia
  Arms: Spinal block

SUMMARY:
There will be compared the postoperative analgesic effect of infiltration or spinal block for hemorrhoidectomy

DETAILED DESCRIPTION:
This is a prospective, randomized study, including 40 patients between 18 and 60 years, of both genders, ASA 1 or 2.

Patients in group 1 (n = 20) will be submitted to spinal block and group 2 (n = 20) to infiltration. The spinal block will be performed with 10 mg of 0.5% bupivacaine. The infiltration will be performed with 10 ml of 0.5% bupivacaine with epinephrine on each side.

Will be evaluated: intensity of pain on a numerical scale from 0 to 10 every 15 minutes, relaxation of the sphincter muscles, intensity of pain after the operation every 30 minutes until reached the criteria for discharge, muscle strength of the lower limbs every 30 minutes, BP, HR, SO2, FR, other items that determine the conditions of discharge (urine output, nausea and vomiting), time to hospital discharge, and duration of analgesia. Adverse effects and complications will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Will be included 50 patients, ASA physical status 1 or 2 undergoing hemorrhoidectomy after approval by the Ethics Committee and signed Consent Form

Exclusion Criteria:

* There will be excluded patients with associated diseases (fistula, fissure), infection at the puncture site, using anticoagulants or analgesics (up to 2 weeks before the procedure) and pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 24 hours
  Numerical score

SECONDARY OUTCOMES:
Time to discharge | 24 hours

OTHER OUTCOMES:
Duration of motor blockade | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rioko K Sakata, PhD, Principal Investigator — Universidade Federal de São Paulo
Locations (1):
- Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No